CLINICAL TRIAL: NCT05904093
Title: A Phase I Study to Evaluate the Safety and Tolerability of Escalating Doses of Fostamatinib in Subjects With Stable Sickle Cell Disease
Brief Title: Study to Evaluate the Safety and Tolerability of Escalating Doses of Fostamatinib in Subjects With Stable Sickle Cell Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10001619; 001619-H
Record Dates: First submitted 2023-06-13; First posted 2023-06-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Sickle Cell Disease; Hb-SS Disease; Hemoglobin S; Disease Sickle Cell Anemia; Sickle Cell Disorders; Hemoglobin Beta Thalassemia Disease
Keywords: Sickle Cell; Tyrosine Kinase Inhibitor; Fostamatinib
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait | interventions — fostamatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fostamatinib in participants with Sickle Cell Disease (Experimental): Participants with Sickle Cell Disease will receive Fostamatinib which will be administered orally, at a dose of 100 mg twice a day for 14 days and if tolerated, will be escalated to a dose of 150 mg, taken orally, twice a day for 28 days (total 42 days).
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib will be administered orally, at a dose of 100 mg twice a day for 14 days and if tolerated, will be escalated to a dose of 150 mg, orally, twice a day for 28 days (total 42 days).

SUMMARY:
Background:

Sickle cell disease (SCD) is a genetic disease that causes the body to produce abnormal ( sickled ) red blood cells. SCD can cause anemia and life-threatening complications in the lungs, heart, kidney, and nerves. People with SCD are also at increased risk of forming blood clots in the veins and lungs, but the standard treatments for these clots can cause increased bleeding in people with SCD. Better treatments are needed.

Objective:

To test a drug (fostamatinib) in people with SCD.

Eligibility:

People aged 18 to 65 with SCD.

Design:

Participants will have 6 clinic visits over 12 weeks. Each visit will be 2 to 3 hours.

Participants will be screened. They will have a physical exam with blood tests. They will tell the researchers about the medications they take.

Fostamatinib is a tablet taken by mouth. Participants will take the drug at home, twice a day, for up to 6 weeks.

Participants will have a clinic visit every 2 weeks while they are taking the drug. At each visit they will have a physical exam with blood tests. They will talk about any side effects the drug may be causing. If they are tolerating the drug well after the first 2 weeks, they may begin taking a higher dose.

Participants will have a final visit 4 weeks after they stop taking the drug. They will have a physical exam and blood tests; they will be checked for any side effects of the drug.

DETAILED DESCRIPTION:
Study Description: The overall objective of this study is to assess the clinical safety and tolerability of fostamatinib in subjects with stable sickle cell disease (SCD). Subjects enrolled will receive fostamatinib 100 mg orally twice daily (BID) for 2 weeks then escalate to 150 mg orally BID for an additional four weeks. Throughout the course of the study subjects will be monitored for signs and symptoms of adverse events. The effect of fostamatinib on laboratory biomarkers of thromboinflammatory activity and red blood cell metabolism will be studied at specified timepoints.

Objectives:

Primary Objective:

To assess the clinical safety and tolerability of fostamatinib, a tyrosine kinase inhibitor with demonstrated activity against spleen tyrosine kinase (Syk), in subjects with stable SCD.

Secondary Objectives:

To assess the pharmacokinetics of fostamatinib in SCD and correlate drug exposure to effects on neutrophil, platelet function, and red cell metabolism to evaluate for anti-sickling and anti-inflammatory effects.

Exploratory Objective:

To gain insight into the exposure response and mechanistic effects of fostamatinib mediated Syk inhibition on intracellular signaling.

Endpoints:

Primary Endpoint:

* To evaluate the safety and tolerability of fostamatinib as assessed by:

  -- frequency and severity of adverse events (AEs) from Baseline to Day 70
* Safety endpoints, including:

  * the type, incidence, severity, and relationship to study treatment of AEs and serious adverse events (SAEs) from Baseline to Day 70 -- number of discontinuations due to AEs; from Baseline to Day 70
  * results of clinical laboratory tests over time and change from baseline (e.g., serum chemistry, liver function test, hematology, coagulation)

Secondary Endpoints:

* Studies of platelet activation and aggregation at baseline, Day 14 following agonist exposure at 100 mg BID, and Day 43 following agonist exposure at 150 mg BID of fostamatinib.
* Evaluate anti-sickling effects of fostamatinib through measures of red blood cell (RBC) membrane band3 tyrosine phosphorylation, RBC deformability, anti-sickling kinetics and oxygen affinity (p50)
* Change from baseline in intracellular reactive oxidative species (ROS) in RBCs at different doses of fostamatinib at regular time intervals (baseline, day 14, and day 43).
* Markers of coagulation activation at regular time intervals (baseline, day 14, and day 43) on fostamatinib and change from baseline.
* Determine peak R406 levels and assess correlation of R406 exposure with inhibition of NETosis and its effect on red blood cell membrane band 3 tyrosine phosphorylation and sickling kinetics at baseline, 1 hr, 2 hrs, 4 hrs, and 8 hrs post dosing (100 mg BID and 150 mg BID)

Exploratory Endpoints:

* Perform mechanistic studies of intracellular signaling pathways relevant to phosphotyrosine kinase inhibition on Day 14 following agonist exposure at 100 mg BID and Day 43 following agonist exposure at 150 mg BID of fostamatinib.
* Measures of neutrophil activation and neutrophil extracellular trap (NET) formation at baseline and following agonistactivation at 100 mg BID versus 150 mg BID of fostamatinib.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will enroll onto the study and undergo screening. Subjects who do not meet any of the following criteria during screening will not receive the study intervention but will be counted toward study accrual. Screen failures may be rescreened at a later time. In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Have provided signed written informed consent prior to performing any study procedure, including screening procedures.
2. Age between 18-65 years
3. Unequivocal diagnosis of SCA (HbSS or HbSBeta^0) confirmed by hemoglobin electrophoresis performed on patients at least 60 days after a blood transfusion if previously transfused.
4. No transfusion in the 60 days prior to signing consent, or absence of Hb A on hemoglobin analysis (by high-performance liquid chromatography; HPLC)
5. Have adequate organ function, as defined by:

   1. Serum aspartate aminotransferase (AST) <=1.5 x Upper Limit of Normal (ULN) (unless the increased AST is assessed by the Investigator as due to hemolysis) and alanine aminotransferase (ALT) <=1.5 x ULN.
   2. Absolute neutrophil count >=1.5 x 10^9/L.
   3. Hemoglobin >= 7 g/dL
   4. Platelet count >=100 x 10^9/L.
6. If on hydroxyurea, participant must have been on stable dose of hydroxyurea (defined as a stable dose for at least 3 months and inclusive of dose modifications for hematological toxicity per PI discretion) prior to signing consent.
7. For women of reproductive potential, have a negative serum pregnancy test during the screening period. Women of reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion; or who have not been naturally postmenopausal (i.e., who have not menstruated at all for at least the preceding 1 year prior to signing informed consent unrelated to hormonal contraception).
8. For women of reproductive potential as well as men and their partners who are women of reproductive potential, be abstinent as part of their usual lifestyle, or agree to use 2 effective forms of contraception from the time of giving informed consent, during the study, and for 28 days (both men and women) following the last dose of study treatment. An effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, intrauterine or subdermal contraceptive implants, and barrier methods.
9. Be willing to comply with all study procedures for the duration of the study.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pain crisis requiring parenteral treatment within 14 days of signing consent.
2. Have a significant medical condition that confers an unacceptable risk to participating in the study, and/or that could confound the interpretation of the study data. Such significant medical conditions include, but are not limited to the following:

   1. History of neutropenia (benign ethnic neutropenia and/or acquired neutropenia related to drug suppression by hydroxyurea and/or cyclic hematopoiesis are permitted).
   2. History of posterior reversible encephalopathy syndrome (PRES)
   3. History of poorly controlled hypertension (defined as systolic blood pressure >=130 mmHg or average diastolic blood pressure >=90 mmHg based on an average of 3 blood pressure readings despite adequate antihypertensive therapy) unless controlled for >90 days prior to enrollment.
   4. Active viral infection as evidenced by testing positive for hepatitis B surface antigen or hepatitis C virus (HCV) antibody (ab) with signs of active hepatitis B or C virus infection. If the subject is positive for HCV Ab, a reverse transcriptase-polymerase chain reaction test will be conducted. Subjects with hepatitis C may be rescreened after receiving appropriate hepatitis C treatment.
   5. History of drug-induced cholestatic hepatitis.
   6. History of any primary malignancy.
   7. Testing positive for human immunodeficiency virus 1 or 2 Ab with evidence for ongoing active infection (i.e., CD 4 count <400/microliter and viral load >100,000 copies/ml) on antiretroviral therapy.
   8. Current or recent history of psychiatric disorder that, in the opinion of the Investigator or Medical Monitor, could compromise the ability of the subject to cooperate with study visits and procedures.
   9. Are currently enrolled in another therapeutic clinical trial involving ongoing therapy with any investigational or marketed product or placebo.
   10. Use of newly approved SCD therapy (L-glutamine, voxelotor or crizanlizumab) is NOT permitted on this study. Subjects who have received newly approved SCD therapy in the 7 days prior to signing consent will be excluded.
   11. Having had a prior bone marrow or stem cell transplant.
   12. Currently pregnant or lactating.
   13. Currently receiving strong inhibitors of CYP3A4/5 that have not been stopped for >=5 days or a time frame equivalent to 5 half-lives (whichever is longer), or strong inducers of CYP3A4 that have not been stopped for >=28 days or a time frame equivalent to 5 half-lives (whichever is longer), prior to signing consent. SCD patients that are receiving treatment with CYP3A4 substrate drugs, some BCRP substrate drugs (eg. rosuvastatin), and some P-glycoprotein substrate drugs (eg. Digoxin) are excluded from the study.
   14. Currently receiving erythropoiesis stimulating agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
The number of type, incidence, severity and relationship to study treatment of adverse events and serious adverse events | Baseline (Day 0) to End of Study (Day 70)
  The type, incidence, severity, and relationship to study treatment of AEs and serious adverse events (SAEs) from baseline to Day according to CTCAE.

SECONDARY OUTCOMES:
Number of participants that discontinued fostamatinib due to adverse events following CTCAE. | Baseline (Day 0) to End of Study (Day 70)
  Number of participants that discontinued fostamatinib due to adverse events following CTCAE from Baseline (Day 0) to End of Study (Day 70)

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001619-H.html